CLINICAL TRIAL: NCT02270320
Title: Study of School and Graduate Institute of Physical Therapy College of Medicine in Taiwan
Brief Title: Cognitive Effects of Tai Chi Chuan in Healthy Older Adults and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201212161RIND; NSC 102-2410-H-002 -213 -MY2 (Other: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2014-09-09; First posted 2014-10-21 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Alteration of Cognitive Function
Keywords: Tai Chi Chuan; cognitive function; motor function; MRI
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control group will receive a telephone consultation once every two weeks for 12 weeks.
- Physical activity (Active Comparator): Experimental group will receive a 60-minute 24 forms Yang-style Tai Chi Chuan exercise program, three times per week for 12 weeks.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The training is 24 forms Yang-style Tai Chi Chuan exercise, which will perform a 60-minute exercise program, three times per week for 12 weeks.
  Arms: Physical activity

SUMMARY:
Background: Promotion of cognitive functions of middle aged and older adults and prevention of dementia are important issues in the aging society. In recent years, studies have shown that Tai Chi Chuan (TCC) exercise can improve cognitive functions in healthy middle-aged and older adults, but not studies have investigated the neural mechanisms. Therefore, the purposes of this research project are: (1) to investigate the effects of TCC exercise intervention on improving cognitive functions and motor functions in healthy middle-aged and older adults; (2) to investigate the effects of TCC intervention on improving the integrity of frontostriatal fiber tracts, and areas and intensity of brain activation while performing a switching task in healthy middle-aged and older adults.

Methods: This project used the assessor-blind and randomized control clinical trial design. A total of 60 healthy middle-aged and older adults will be recruited, randomly allocated to two groups: experimental and control groups. Experimental group will receive a 60-minute exercise program, three times per week for 12 weeks. Control group will receive a telephone consultation once every two weeks for 12 weeks. All participants will receive clinical neuropsychological tests, Cambridge Neuropsychological Test Automated Battery tests, motor function tests, diffusion spectrum MR imaging, and functional MRI experiments before intervention, and at the end of intervention to realize the changes of cognitive function, motor function, integrity of neural tracts, and intensity and regions of functional activation while doing switching task of executive function in order to understand the cognitive effects and the neural mechanisms of TCC.

DETAILED DESCRIPTION:
Background: Promotion of cognitive functions of middle aged and older adults and prevention of dementia are important issues in the aging society. In recent years, studies have shown that Tai Chi Chuan (TCC) exercise can improve cognitive functions in healthy middle-aged and older adults, but not studies have investigated the neural mechanisms. Therefore, the purposes of this research project are: (1) to investigate the effects of TCC exercise intervention on improving cognitive functions and motor functions in healthy middle-aged and older adults; (2) to investigate the effects of TCC intervention on improving the integrity of frontostriatal fiber tracts, and areas and intensity of brain activation while performing a switching task in healthy middle-aged and older adults.

Methods: This project used the assessor-blind and randomized control clinical trial design. A total of 60 healthy middle-aged and older adults will be recruited, randomly allocated to two groups: experimental and control groups. Experimental group will receive a 60-minute exercise program, three times per week for 12 weeks. Control group will receive a telephone consultation once every two weeks for 12 weeks. All participants will receive clinical neuropsychological tests, Cambridge Neuropsychological Test Automated Battery tests, motor function tests, diffusion spectrum MR imaging, and functional MRI experiments before intervention, and at the end of intervention to realize the changes of cognitive function, motor function, integrity of neural tracts, and intensity and regions of functional activation while doing switching task of executive function in order to understand the cognitive effects and the neural mechanisms of TCC.

ELIGIBILITY:
Inclusion Criteria:

* age range between 50 - 85 years old.
* education level > 6 years or can read and speak Chinese
* Montreal Cognitive Assessment Taiwan version (MoCA) score >= 26
* Clinical Dementia Rating (CDR) score = 0
* right dominant hand

Exclusion Criteria:

* any neurological diseases, ex stroke, Parkinson's disease, trauma, epilepsy
* cardiac disease, cardiac infarction, angina, uncontrolled hypertension
* spiritual disease, anxiety or depression (Geriatric Depression Scale 15-item short-form score >= 8)
* Daily ability need helps (instrumental activities of daily living, IADL has one item score= 0 or 1)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
General cognitive function | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Cognitive score on Montreal Cognitive Assessment Taiwan version (MoCA) and Clinical Dementia Rating (CDR).
Executive function | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Completed time (seconds) on Color Trail Test- Part 1& 2, and number of errors from executive function task on Cambridge Neuropsychological Test Automated Battery (CANTAB).
Motor strength | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Upper and lower limbs' muscle strength (kg) on handheld dynamometer, grip test, and to test lower limb strength by measuring the completed times in 30 seconds, chair rise test.
Flexibility | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Flexibility score (cm) on scratch test, chair sit and reach test.
Balance | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Balance time (seconds) on eyes opened one-leg stance test.
Coordination | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Coordination time (seconds) on four square step test and "Timed Up and Go" test
Endurance | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Walking distance (meters) on six-minute walking test.
Physical activity level | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Physical activity score on "Physical Activity Scale for the Elderly" questionnaire.
Memory function | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Memory score on Cambridge Neuropsychological Test Automated Battery (CANTAB).

SECONDARY OUTCOMES:
Brain functional activation | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Brain MR images were obtained with a 3T Siemens (Erlangen, Germany) whole-body MRI scanner. A Siemens 32-channel head array coil was used as a receiver. Functional MRI (fMRI) was acquired using a BOLD-weighted gradient-echo echoplanar image sequence (EPI) ( TR/TE=2000/24 ms, field of view= 192 mm, voxel dimensions 3 x 3 x 4 mm, matrix= 64 x 64, slice thickness= 4 mm, flip angle 90°), and 34 slices will be obtained with anterior-posterior phase encoding direction and covering the whole brain. The fMRI paradigm was the event-related designed switching task by E-prime 2.0. The fMRI imaging data processing and analysis were accomplished using SPM8 (Wellcome Department of Imaging Neuroscience). Statistical parametric maps of the t statistic, SPM{t}, were obtained with the threshold of p< 0.001 uncorrected. The brain functional activation results will be presented by the p value and the magnitude of Blood-oxygen-level dependent (BOLD) intensity.
Brain structural integrity | This outcome will be assessed at baseline and up to 12 weeks exercise or control intervention.
  Structural MRI was measured by T1, T2, and diffusion spectrum imaging (DSI). DSI will be performed to reconstruct tractography of the neural tracts. The DSI data was acquired by using a pulsed-gradient spin-echo diffusion EPI. The maximum diffusion sensitivity b value=4000 s/mm2, TR/TE=9600/130 ms, FOV=200 mm, and thickness=2.5 mm. Approximately 56 transaxial slices will be acquired encompassing the whole brain. The general fractional anisotropy (GFA) values, a quantitative index derived from the orientation distribution function to indicate diffusion anisotropy, were calculated at each voxel, The reconstruction of the tracts tractography was performed by using DSI Studio software. The integrity of these neural tracts will be presented by GFA value.

OTHER OUTCOMES:
Handness | This outcome will be assessed at baseline.
  Handness score on "Edinburgh Handedness Inventory" questionnaire.
Footness | This outcome will be assessed at baseline.
  Footless score on "Waterloo Footedness Questionnaire".
Emotion | This outcome will be assessed at baseline.
  Depression score on "Geriatric Depression Scale 15-item short-form".
Basic physical function | This outcome will be assessed at baseline.
  Basic physical score on " instrumental activities of daily living" questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Study Chair — School and Graduate Institute of Physical Therapy College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan